CLINICAL TRIAL: NCT06294223
Title: Investigation of the Correlation Between Upper Extremity Fatigue Level and Muscle Oxygenation
Brief Title: Upper Extremity and Muscle Oxygenation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tuna Sümer, PT, Saglik Bilimleri Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SaglikBilU
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Near-infrared Spectroscopy; Muscle Oxygenation
Keywords: Near-infrared Spectroscopy; Resistance Exercise; Exercise Intensity; Muscle Oxygenation; Muscle Activation
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement of Upper Extremity Muscle Oxygenation (Experimental): Measuring muscle oxygenation with fatigue protocol.
  Interventions: Device: Exercise follow up with near-infrared spectroscopy

INTERVENTIONS:
Device: Exercise follow up with near-infrared spectroscopy — Exercises will be followed by near-infrared spectroscopy. Fatigue protocol will be applied.

SUMMARY:
The aim of this study was to measure the acute change in oxygen saturation of skeletal muscle during resistance exercise in the upper extremity using near-infrared spectroscopy.

DETAILED DESCRIPTION:
Our study aims to determine the acute oxygen response in the upper extremity muscles against a resistance exercise fatigue protocol, in order to demonstrate the effect of muscle oxygenation levels on the occurrence of symptoms such as fatigue in upper extremity use, and to provide reference information for the development of exercise programs.

It is known that resistance exercise increases resting energy expenditure and promotes fat oxidation for weight loss. Changes in cardiopulmonary function that occur in chronic diseases reduce oxygen uptake and decrease energy production, leading to increased fatigue. Resistance exercises in chronic diseases can regulate an individual's energy production capacity.

The main objective of our study is to investigate the effect of muscle oxygenation levels on the occurrence of symptoms such as fatigue by determining the oxygen response in the upper extremity muscles based on a resistance exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being over 18 years old
* Having a Body Mass Index (BMI) value between 23-30 kg/m2
* Absence of comorbid disease of the orthopedic, neurological, cardiopulmonery system

Exclusion Criteria:

* Smoking / alcohol use
* Presence of orthopedic disease effecting the upper extremity or previous surgery
* Presence of cardiopulmonery disease that prevents exercise
* Participants who performed resistance exercise regulary for more than 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Determination of Blood Pressure | Measurement will be made before and immediately after exercise.
  Systolic/diastolic blood pressure will be determined with a digital blood pressure monitor and will be recorded in mmHg. Measurements will be taken via the right brachial artery in a comfortable position.
Saturation Measurement | Measurement will be made before and immediately after exercise.
  Oxygen saturation will be measured with a pulse oximeter device and recorded on the form.
Muscle Oxygenation Measurement | Baseline.
  MOXY Pro (Moxy 3, Firmware 1.1 Hutchinson MN, USA), a near-infrared spectroscopy device, will be used to measure the muscle oxygen rate (SmO2) and total hemoglobin amount (tHb) of the biceps brachii muscle.
Determination of Heart Rate | Measurement will be made before and immediately after exercise.
  Heart rate will be determined with a digital blood pressure monitor and will be recorded in BPM.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, Ass. Prof., Study Director — Saglik Bilimleri Universitesi; Mehmet Burak Uyaroğlu, Pt.PhD(c), Principal Investigator — Saglik Bilimleri Universitesi; Tuna Sümer, PT, Study Chair — Saglik Bilimleri Universitesi; Melisa Eren, PT, Study Chair — Saglik Bilimleri Universitesi; Ceren Balıkcı, PT, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No